CLINICAL TRIAL: NCT00270231
Title: Pharmacogenetic Investigation of Naltrexone
Brief Title: Effects of Naltrexone on Nicotine Reinforcement
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: 800810; R01DA017555 (NIH)
Record Dates: First submitted 2005-12-23; First posted 2005-12-26 (Estimated); Results first posted 2013-12-10 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-11

CONDITIONS: Tobacco Dependence
Keywords: within-subjects, crossover, laboratory study; Naltrexone vs. Placebo
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Naltrexone (Active Comparator): All participants took naltrexone during one of the two 4-day study medication periods. Both 4-day study medication periods were randomized and counterbalanced between naltrexone and placebo; all study medication periods were separated by a 5-7 day washout period.
  Dosing of the naltrexone was the same for all participants: Day 1: 12.5mg, Day 2: 25mg, Days 3 and 4: 50mg.
  Interventions: Drug: Naltrexone
- Placebo (Placebo Comparator): All participants took a placebo (sugar pill) during one of the two 4-day study medication periods. Both 4-day study medication periods were randomized and counterbalanced between naltrexone and placebo.
  Placebo capsules matched the naltrexone in color, weight and inactive ingredients. The only difference the lack of active naltrexone in each capsule.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone — All participants took naltrexone during one of the two 4-day study medication periods. Both 4-day study medication periods were randomized and counterbalanced between naltrexone and placebo; all study medication periods were separated by a 5-7 day washout period.
  Dosing of the naltrexone was the same for all participants: Day 1: 12.5mg, Day 2: 25mg, Days 3 and 4: 50mg.
  Other Names: Revia or Trexan
  Arms: Naltrexone
Drug: Placebo — All participants took a placebo (sugar pill) during one of the two 4-day study medication periods. Both 4-day study medication periods were randomized and counterbalanced between naltrexone and placebo.
  Placebo capsules matched the naltrexone in color, weight and inactive ingredients. The only difference the lack of active naltrexone in each capsule.
  Other Names: Sugar pill; inactive medication
  Arms: Placebo

SUMMARY:
Despite preclinical evidence supporting the role of the endogenous opioid system in the reinforcing effects of nicotine, the efficacy of the opioid antagonist naltrexone (NTX) as a tobacco dependence treatment remains unresolved. Research is needed to identify those smokers for whom NTX will have the strongest beneficial effects on smoking behavior.

The research bridges existing knowledge of genetic, pharmacologic, and behavioral responses to nicotine, and translates this knowledge to treatment for tobacco dependence. The immediate goal was to test whether genetic variation in the mu-opioid receptor gene predicts the effects of naltrexone (NTX) on nicotine reinforcement.

DETAILED DESCRIPTION:
The study was a within-subject double-blind study of the effects of naltrexone versus placebo on the reinforcing value of nicotine, using a validated cigarette choice paradigm. A key question was whether smokers differ in their responses based on the mu opioid receptor gene (OPRM1) Asn40Asp (A118G) variant.

Following informed consent, 64 smokers were enrolled in the study. Of these, 60 completed two 4-day study phases interspersed with a 5-7 day washout phase. Baseline statistics are provided for the 64 smokers who enrolled.

Each 4-day study phase included a 3-day drug run-up and monitoring phase, then on the 4th day participants came to our Biobehavioral Lab (BBL) where they took their final 50mg of study medication and completed a cigarette choice paradigm. Following a washout phase, the 4-day sequence will be repeated with the alternative study medication. The order of study medication was randomized and counterbalanced between subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be greater than or equal to 18 years
2. Based on the medical history, physical and laboratory examination, female subjects must:

   1. Agree in consent to practice effective contraception during study, be status post-bilateral tubal litigation or be post-menopausal.
   2. Not be pregnant, nursing, or planning pregnancy
3. Based upon self-report, subjects must smoke greater than or equal to 10 non-menthol cigarettes per day
4. Because the OPRM1 variant is common (25-30%) in persons of European ancestry, but very rare in other ethnic groups (e.g., 2-9% of African Americans) it is not scientifically justified to include members of other ethnic groups. Therefore, only persons of European ancestry will be recruited.
5. Following orientation by the research staff, subjects must sign written informed consent and HIPAA form.

Exclusion Criteria:

1. Current diagnosis of kidney disease or history of renal function impairment (unless they have recent kidney function tests (within last 3 months) and approval of their primary physician to participate in the study.)
2. Women who are pregnant, planning a pregnancy, or lactating
3. Current alcohol use > 25 standard drinks/week (this is because NTX is used to treat alcohol dependence, and effects of NTX on alcohol consumption in alcohol dependent subjects could have indirect effects on cigarette consumption).
4. Current medical problems for which NTX is contraindicated including: active hepatitis (Liver Function Tests 3 times the Upper Limit of Normal).
5. History of opiate dependence (prescription drug or illicit use).
6. History of or current Diagnostic and Statistical Manual of Mental Disorders (Version IV) (DSM IV) substance use disorders (abuse or dependence involving alcohol, cocaine, stimulants, or benzodiazepines)
7. Diagnosis of bulimia and/or anorexia nervosa in the last year
8. Current or past use (with in past 12 months) of any medications containing NTX (e.g., Revia, Trexan), allergy to NTX
9. Concomitant medications (e.g., monoamine oxidase inhibitors or benzodiazepines within past 14 days, antipsychotics, antidepressants, theophylline, systemic steroids, over-the-counter stimulants and anorectics)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2004-03; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caryn Lerman, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- Tobacco Use Research Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Ray R, Jepson C, Wileyto P, Patterson F, Strasser AA, Rukstalis M, Perkins K, Blendy J, Lerman C. CREB1 haplotypes and the relative reinforcing value of nicotine. Mol Psychiatry. 2007 Jul;12(7):615-7. doi: 10.1038/sj.mp.4002002. No abstract available. PMID 17592483
- [Result] Ray R, Jepson C, Patterson F, Strasser A, Rukstalis M, Perkins K, Lynch KG, O'Malley S, Berrettini WH, Lerman C. Association of OPRM1 A118G variant with the relative reinforcing value of nicotine. Psychopharmacology (Berl). 2006 Oct;188(3):355-63. doi: 10.1007/s00213-006-0504-2. Epub 2006 Sep 8. PMID 16960700

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from March 2004 to August 2005. All subject sessions occurred at the Tobacco Use Research Center's lab, the Biobehavioral Lab (BBL), at the University of Pennsylvania.
Pre-assignment Details: The primary genotype of interest was the functional mu opioid receptor (OPRM1). Smokers with the Asp40 variant (A/G or G/G genotypes; about 27% of smokers) were oversampled, relative to those with the more common Asn40 variant (A/A genotype; 73% of smokers), in order to have an equal number of participants in each genotype group.
Groups:
- Naltrexone, Then Placebo: These participants took active naltrexone during their first 4-day study period. The dosing for naltrexone was the same for all participants. Day 1 = 12.5mg, Day 2 = 25mg, Days 3 & 4 = 50mg.
  They received placebo (sugar pill) during the second 4-day study period.
- Placebo, Then Naltrexone: These participants took placebo (sugar pill) during their first 4-day study period.
  They received active naltrexone during the second 4-day study period. The dosing for naltrexone was the same for all participants. Day 1 = 12.5mg, Day 2 = 25mg, Days 3 & 4 = 50mg.
Period: First Intervention
Arm/Group | Naltrexone, Then Placebo | Placebo, Then Naltrexone
Started | 32 | 32
Completed | 31 | 31
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1
Period: Washout Period
Arm/Group | Naltrexone, Then Placebo | Placebo, Then Naltrexone
Started | 31 | 31
Completed | 30 | 31
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Second Intervention
Arm/Group | Naltrexone, Then Placebo | Placebo, Then Naltrexone
Started | 30 | 31
Completed | 30 | 30
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes subjects with both OPRM1 genotypes (Asp40 (A/G or G/G allele vs. Asn40 (A/A) allele) who started Intervention Period 1.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 59
  >=65 years | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 43.2 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 38
Region of Enrollment [Number; unit: participants]
  United States | 64

OUTCOME MEASURES:

1. Primary Outcome: Number of Nicotine Cigarette Choices Taken During the Cigarette Choice Procedure.
Description: On day 4 of each study medication period, participants completed a cigarette choice procedure where the subject is asked to take 4 puffs from a nicotinized (nicotine-containing) or a denicotinized (no nicotine) cigarette every 30 minutes for 2 hours (maximum of 24 puffs). The outcome variable is the number of nicotine cigarette choices or puffs out of 24 total puffs during these cigarette choice procedures.
  Subjects who had the A/A genotype took an average of 18.5 puffs from the nicotine-containing cigarettes. Subjects with the A/G or G/G genotypes took an average of 16.2 puffs from the nicotine-containing cigarettes.
Time Frame: 2 hours
Population: Participants were analyzed with respect to genotype regardless of intervention.
Measure: Mean (Standard Deviation); unit: Number of Nicotine Cigarette Puffs Taken
Groups:
- OPRM1 Genotype - A/A: Participants who have the Asn40 OPRM1=A/A
- OPRM1 Genotype - A/G or G/G: Participants who have the Asp40 OPRM1=A/G or G/G
Arm/Group | OPRM1 Genotype - A/A | OPRM1 Genotype - A/G or G/G
Number analyzed (Participants) | 30 | 30
Number of Nicotine Cigarette Puffs Taken | 18.5 (4.2) | 16.2 (6.2)

ADVERSE EVENTS:
Groups:
- Naltrexone Only: Active medication recipients (Naltrexone taken for 4 days).
- Placebo Only: Placebo (sugar pill) recipients (taken for four days).
Arm/Group | Naltrexone Only | Placebo Only
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/64
Other Adverse Events (participants affected / at risk) | 0/64 | 0/64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No